CLINICAL TRIAL: NCT02529618
Title: Implementation of iDETECT for Field Triage of mTBI in Football Players
Brief Title: Field Implementation of iDETECT
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: National Football League (Other)
Responsible Party: Principal Investigator, Tamara Espinoza, MD, Assistant Professor, Emory University
Other Study IDs: IRB00082102
Record Dates: First submitted 2015-08-19; First posted 2015-08-20 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-03

CONDITIONS: Concussion; Brain Trauma
MeSH Terms: conditions — Brain Concussion; Brain Injuries, Traumatic | interventions — Drug Delivery Systems

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Football Athlete Group: All football athlete participants in this arm will take the integrated Display Enhanced Testing for Cognitive Impairment and mild traumatic brain injury (iDETECT) test. Participants who sustain a concussion during the football season will complete the iDETECT test and a standing balance test (BESS assessment) four times after injury. Participants in this arm are eligible to receive the Riddell High Impact Technology (HIT) System or the i1 Biometrics Vector Mouth Guard.
  NOTE: Football athletes who sustain a concussion during the football season will be evaluated and managed according to standard concussion screening and return-to-play (RTP) protocols. Performance on iDETECT or other study related tasks will NOT be used to make diagnosis, management, or return to play decisions. Study staff will not assist with or influence diagnosis, management, or return-to-play decision making by teams' medical personnel.
  Interventions: Device: integrated Display Enhanced Testing for Cognitive Impairment and mild traumatic brain injury (iDETECT); Device: Riddell High Impact Technology (HIT) System; Device: i1 Biometrics Vector Mouth Guard
- Non-Collision Sport Athlete Group: Non-collision sport athletes who are active in a school's Fall athletic program will be take the integrated Display Enhanced Testing for Cognitive Impairment and mild traumatic brain injury (iDETECT) test, standing balance test (BESS assessment), and complete a questionnaire at the beginning of the sport season. Participants will be asked to take the iDETCT test up to 5 more times during the season. Participants who sustain a concussion during the athletic season will be asked to take additional iDETECT tests four times after the injury.
  NOTE: Non-collision sport athletes who sustain a concussion during the season will be evaluated and managed according to standard concussion screening and return-to-play (RTP) protocols. Performance on iDETECT or other study related tasks will NOT be used to make diagnosis, management, or return to play decisions. Study staff will not assist with or influence diagnosis, management, or return-to-play decision making by teams' medical personnel.
  Interventions: Device: integrated Display Enhanced Testing for Cognitive Impairment and mild traumatic brain injury (iDETECT)

INTERVENTIONS:
Device: integrated Display Enhanced Testing for Cognitive Impairment and mild traumatic brain injury (iDETECT) — iDETECT offers an open platform for an evaluation of cognitive, balance, and oculomotor performance after mild traumatic brain injury (mTBI). It is a rugged, portable, neurocognitive assessment tool designed specifically for use in field and triage settings for the rapid evaluation of functional neurologic impairment after potential concussive injury.
Device: Riddell High Impact Technology (HIT) System — The Riddell HIT system incorporates six acceleration sensors into standard football helmets worn during practice and game play. A computerized sideline system captures information on linear and rotational acceleration, as well as magnitude, duration, and location of impact for each player
  Groups: Football Athlete Group
Device: i1 Biometrics Vector Mouth Guard — The i1 Biometrics Vector Mouth Guard is an impact intelligence system that contains a collection of impact sensing mouth guards, housing accelerometer and gyroscope technology that allows real-time collection and storage of biomechanical impact data. Sensors in the mouth guard communicate directly with a sideline assessment base station and allows for immediate assessment and evaluation of hit exposure.
  Groups: Football Athlete Group

SUMMARY:
The purpose of this study is to assess a new screening tool for sideline evaluation of concussion injuries in athletes. iDETECT is a new technology that combines several elements of recommended concussion screening tools into a single, portable device.

DETAILED DESCRIPTION:
The goal of the research is to evaluate the use of a multimodal platform (iDETECT) for immediate post-injury neuropsychological, balance and oculomotor assessment, and to evaluate the iDETECT platform as a return-to-play assessment tool during the post injury management period following concussion.

ELIGIBILITY:
Inclusion Criteria:

* Athletes participating in the Fall 2015 high school season
* Aged 14 years or older
* No concussion injuries within prior 2 months
* Provide signed and data consent and/or assent form(s)

Exclusion Criteria:

* Non-English speaking
* History of seizures or prior brain surgery (excluding facial and TM surgery)
* Concussion within last 2 months
* Poor Effort on baseline iDETECT test

Non-Collision Sport Group

* current concussion or history of current concussion during the Fall 2015 athletic season

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: iDETECT will be used to assess neuro-functional outcomes known to be impaired after mTBI in competitive high school athletic teams over a standard season.
  Eligible participants include: a) all football athletes at participating high schools; b) all non-football athletes who sustain a concussion during the Fall 2015 season; c) interested non-collision sport athletes without a concussion (to serve at controls).
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2015-08; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC) for iDetect total score of neuropsychological assessment (NP) compared to the trainer's determination of clinical concussion | Baseline, throughout duration of sport season (an expected average of 4 months)
  The area under the receiver operator characteristic (ROC) curve (the concordance index) for total score of NP will be computed and compared with the trainer's determination of clinical concussion to find out if iDETECT is as accurate in diagnosing concussion.
Area under the curve (AUC) for iDetect NP total score compared to the Immediate Post-Concussion Assessment and Cognitive Testing (ImPACT) score | Baseline, throughout duration of sport season (an expected average of 4 months)
  The area under the receiver operator characteristic (ROC) curve (the concordance index) for total score of NP will be computed and compared to the ImPACT score to find out if iDETECT is as accurate in diagnosing concussion.
Area under the curve (AUC) for iDetect NP response time to stimuli compared to the trainer's determination of clinical concussion | Baseline, throughout duration of sport season (an expected average of 4 months)
  The area under the receiver operator characteristic (ROC) curve (the concordance index) for NP response will be computed and compared trainer's determination of clinical concussion to find out if iDETECT is as accurate in diagnosing concussion.
Area under the curve (AUC) for iDetect NP response time to stimuli compared to Immediate Post-Concussion Assessment and Cognitive Testing (ImPACT) score | Baseline, throughout duration of sport season (an expected average of 4 months)
  The area under the receiver operator characteristic (ROC) curve (the concordance index) for NP response will be computed and compared the ImPACT score to find out if iDETECT is as accurate in diagnosing concussion.
Area under the curve (AUC) for iDETECT total score compared to final clinical determination of concussion | Baseline, throughout duration of sport season (an expected average of 4 months)
  The area under the receiver operator characteristic (ROC) curve (the concordance index) for iDETECT total score will be compared to the trainer's final clinical determination of concussion.
Area under the curve (AUC) for iDETECT total score compared to the Sport Concussion Assessment Tool (SCAT3) | Baseline, throughout duration of sport season (an expected average of 4 months)
  The area under the receiver operator characteristic (ROC) curve (the concordance index) for iDETECT total score will be compared to the SCAT 3 score. SCAT3 is a standardized tool for evaluating injured athletes for concussion.

SECONDARY OUTCOMES:
Area under the curve (AUC) for iDETECT Non-postural Balance/Sensory Integration (SI) battery time to balance compared to trainer's determination of clinical concussion | Baseline, throughout duration of sport season (an expected average of 4 months)
  The area under the receiver operator characteristic (ROC) curve (the concordance index) for SI battery time will be computed and compared to the trainer's determination of clinical concussion to find out if iDETECT is as accurate in diagnosing concussion.
Area under the curve (AUC) for iDETECT Non-postural Balance/Sensory Integration (SI) battery time to balance compared to Balance Error Scoring System (BESS) score | Baseline, throughout duration of sport season (an expected average of 4 months)
  The area under the receiver operator characteristic (ROC) curve (the concordance index) for SI battery time will be computed and compared to BESS score to find out if iDETECT is as accurate in diagnosing concussion.The SI battery requires participants to utilize primary sensory inputs to assess the state of a virtual balance beam displayed within the iDETECT visor immersive environment without standing.
Area under the curve (AUC) for iDETECT Non-postural Balance/Sensory Integration (SI) battery number of overshoots compared to BESS score | Baseline, throughout duration of sport season (an expected average of 4 months)
  The area under the receiver operator characteristic (ROC) curve (the concordance index) for SI battery number of overshoots will be computed and compared to the BESS score to find out if iDETECT is as accurate in diagnosing concussion.
Area under the curve (AUC) for iDETECT Vestibular and Oculomotor (VO) battery angle difference in target motion prediction compared to trainer's determination of clinical concussion | Baseline, throughout duration of sport season (an expected average of 4 months)
  The area under the receiver operator characteristic (ROC) curve (the concordance index) for VO battery angle distance in target motion prediction will be computed and compared to the trainer's determination of clinical concussion to find out if iDETECT is as accurate in diagnosing concussion.
Area under the curve (AUC) for iDETECT Vestibular and Oculomotor (VO) battery angle difference in target motion prediction compared to King-Devick score (time and number of errors) | Baseline, throughout duration of sport season (an expected average of 4 months)
  The area under the receiver operator characteristic (ROC) curve (the concordance index) will be computed and compared to the King-Devick score (time and number of errors).
Area under the curve (AUC) for iDETECT Vestibular and Oculomotor (VO) battery angle difference in target motion interefence compared to trainer's determination of clinical concussion | Baseline, throughout duration of sport season (an expected average of 4 months)
  The area under the receiver operator characteristic (ROC) curve (the concordance index) for VO battery angle difference in target motion interference will be computed and compared to the trainer's determination of clinical concussion to find out if iDETECT is as accurate in diagnosing concussion.
Area under the curve (AUC) for iDETECT Vestibular and Oculomotor (VO) battery angle difference in target motion interefence compared to King-Devick score (time and number of errors) | Baseline, throughout duration of sport season (an expected average of 4 months)
  The area under the receiver operator characteristic (ROC) curve (the concordance index) for VO battery angle difference in target motion interference will be computed and compared to the to King-Devick score (time and number of errors) to find out if iDETECT is as accurate in diagnosing concussion.
Change in iDETECT total score from baseline to time of injury | Baseline, time of concussion
  Difference in iDETECT total score from baseline to time of concussion will be used to calculate the degree of discrimination in concussed athletes.
Change in iDETECT total score from baseline to end of season to assess subconcussion | Baseline, end of sport season (an expected average of 4 months)
  Mean scores between cases and controls will be compared on iDETECT. Change is defined as the difference in scores from baseline to the end of the season.
Change in Sport Concussion Assessment Tool 3 (SCAT3) total score from baseline to end of season to assess subconcussion | Baseline, end of sport season (an expected average of 4 months)
  Mean scores between cases and controls will be compared using the SCAT3. Change is defined as the difference in scores from baseline to the end of the season.
iDETECT word recall score post injury | 3 days post injury (3 minutes)
  Subjects are asked to remember a group of 12 words displayed one at a time. They are then shown 24 words and asked to respond 'YES' for a word in the original list and 'NO' for a word that was not in the original list. Subjects are scored on the number of words they correctly remember being on the list.
Change in iDETECT mean word recall score post injury, 10 days | 3 days post injury (3 minutes), 10 days post injury (3 minutes)
  Subjects are asked to remember a group of 12 words displayed one at a time. They are then shown 24 words and asked to respond 'YES' for a word in the original list and 'NO' for a word that was not in the original list. Subjects are scored on the number of words they correctly remember being on the list. Change is defined as the difference in scores from 3 days post injury to 10 days post injury.
Change in iDETECT mean word recall score post injury, 30 days | 10 days post injury (3 minutes), 30 days post injury (3 minutes)
  Subjects are asked to remember a group of 12 words displayed one at a time. They are then shown 24 words and asked to respond 'YES' for a word in the original list and 'NO' for a word that was not in the original list. Subjects are scored on the number of words they correctly remember being on the list. Change is defined as the difference in scores from 10 days post injury to 30 days post injury.
iDETECT shapes test score post injury | 3 days post injury (2 minutes)
  Subjects are presented a shape stimulus with 3 characteristics: shape, color, and crosshatch orientation and asked to remember the object. The subject selects the correct shape with 'YES' and each incorrect shape with 'NO'. Score is calculated by correctly selecting the shape.
Change in iDETECT mean shapes test score post injury, 10 days | 3 days post injury (2 minutes), 10 days post injury (2 minutes)
  Subjects are presented a shape stimulus with 3 characteristics: shape, color, and crosshatch orientation and asked to remember the object. The subject selects the correct shape with 'YES' and each incorrect shape with 'NO'. Score is calculated by correctly selecting the shape. Change is defined as the difference in scores from 3 days post injury to 10 days post injury.
Change in iDETECT mean shapes test score post injury, 30 days | 10 days post injury (3 minutes), 30 days post injury (3 minutes)
  Subjects are presented a shape stimulus with 3 characteristics: shape, color, and crosshatch orientation and asked to remember the object. The subject selects the correct shape with 'YES' and each incorrect shape with 'NO'. Score is calculated by correctly selecting the shape. Change is defined as the difference in scores from 10 days post injury to 30 days post injury.
iDETECT arrows test score post injury | 3 days post injury (2 minutes)
  Subjects are asked to respond to an arrow with 2 characteristics: orientation and color. If the arrow is blue, they select the side that the arrow is pointing. If the arrow is red, they select the side opposite from where it is pointing. Score is calculated by the number of correct responses.
Change in iDETECT mean arrows test score post injury, 10 days | 3 days post injury (2 minutes), 10 days post injury (2 minutes)
  Subjects are asked to respond to an arrow with 2 characteristics: orientation and color. If the arrow is blue, they select the side that the arrow is pointing. If the arrow is red, they select the side opposite from where it is pointing. Score is calculated by the number of correct responses. Change is defined as the difference in scores from 3 days post injury to 10 days post injury.
Change in iDETECT mean arrows test score post injury, 30 days | 10 days post injury (2 minutes), 30 days post injury (2 minutes)
  Subjects are asked to respond to an arrow with 2 characteristics: orientation and color. If the arrow is blue, they select the side that the arrow is pointing. If the arrow is red, they select the side opposite from where it is pointing. Score is calculated by the number of correct responses. Change is defined as the difference in scores from 10 days post injury to 30 days post injury.
iDETECT N-BACK (1-back and 2-back) test post injury | 3 days post injury (2 minutes)
  Subjects view a series of faces one at a time and choose if the face has been shown before. The subject selects 'YES' if the face shown is the same as the previous or 'NO' if it is not. Score is calculated by the number of correct responses.
iDETECT Delayed Word Recall Test | 3 days post injury (2 minutes)
  Subjects are asked to recite words from the word recall test after a five minute delay. Score is calculated by the number of words correctly recalled.
Change in iDETECT Delayed Word Recall Test | 3 days post injury (2 minutes), 10 days post injury (2 minutes)
  Subjects are asked to recite words from the word recall test after a five minute delay. Score is calculated by the number of words correctly recalled. Change is defined as the difference in scores from 3 days post injury to 10 days post injury.
Change in iDETECT Delayed Word Recall Test | 10 days post injury (2 minutes), 30 days post injury (2 minutes)
  Subjects are asked to recite words from the word recall test after a five minute delay. Score is calculated by the number of words correctly recalled. Change is defined as the difference in scores from 10 days post injury to 30 days post injury.

CONTACTS AND LOCATIONS:
Overall Officials: Tamara Espinoza, MD, MPH, Principal Investigator — Emory University
Locations (4):
- United States (4):
  - Westminster High School, Atlanta, Georgia
  - Woodward Academy, College Park, Georgia
  - Marietta High School, Marietta, Georgia
  - Blessed Trinity Catholic High School, Roswell, Georgia